CLINICAL TRIAL: NCT06028633
Title: Efficacy and Safety of Albumin-bound Paclitaxel-Lenvatinib-Pembrolizumab in Advanced Nonsquamous NSCLC Patients After Progression to First-line Anti-PD-1/L1 Inhibitor With Platinum-doublet Chemotherapy
Brief Title: Efficacy and Safety of Nab-paclitaxel-Lenvatinib-Pembrolizumab as Second-line Treatment in Advanced NSCLC Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Shikai Wu, professor, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISP61001
Record Dates: First submitted 2023-08-22; First posted 2023-09-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Advanced Non-squamous Non-small-cell Lung Cancer; Recurrent Non-Squamous Non-Small Cell Lung Cancer; Metastatic Non-squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab; lenvatinib; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm I (Experimental): Participants will receive pembrolizumab IV 200 mg D1 every 3 weeks, lenvatinib 8 mg orally every day, albumin-bound paclitaxel IV 100mg/m2 D1, 8 every 3 weeks,until disease progression, intolerable toxicity, investigator decision, or completion of 35 cycles(for pembrolizumab) and 4-6 cycles(for albumin-bound paclitaxel).
  Interventions: Drug: pembrolizumab; Drug: lenvatinib; Drug: albumin-bound paclitaxel

INTERVENTIONS:
Drug: pembrolizumab — pembrolizumab 200mg IV on day 1 for every 3 weeks
  Other Names: Keytruda
Drug: lenvatinib — lenvatinib 8mg taken orally every day
  Other Names: Lenvima
Drug: albumin-bound paclitaxel — albumin-bound paclitaxel IV 100mg/m2 D1, 8 every 3 weeks
  Other Names: nab-paclitaxel; paclitaxel for injection(albumin bound)

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of albumin-bound paclitaxel-lenvatinib-pembrolizumab in advanced nonsquamous NSCLC patients after progression to first-line anti-PD-1/L1 inhibitor with platinum-doublet chemotherapy. All participants will be given with albumin-bound paclitaxel, lenvatinib and pembrolizumab.

ELIGIBILITY:
Inclusion criteria

1. Male/female participants who are at least 18 years of age on the day of signing informed consent (ICF) with histologically confirmed diagnosis of metastatic nonsquamous NSCLC (AJCC Staging Manual, Version 8) will be enrolled in this study.
2. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
3. Male participants are eligible to participate the study if they agree to the following during the intervention period and for at least 180 days after the last dose of study intervention:

   Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR must agree to use contraception unless confirmed to be azoospermia (vasectomized or secondary to medical cause) as:

   A. Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.

   B. Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions is more stringent than the requirements above, the local label requirements are to be followed.

   C. Please note that 7 days after lenvatinib is stopped, if the participant is on pembrolizumab only, no male contraception measures are needed D. Refrain from donating sperm for at least 120 days after the last dose of Lenvatinib.
4. Female participant is eligible to participate if she is not pregnant or not breastfeeding, and at least one of the following conditions applies:

   A. Not a woman of childbearing potential (WOCBP).

   B. A WOCBP who agrees to follow the contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the treatment period and for at least 120 days after the last dose of pembrolizumab or 30 days after the last dose of lenvatinib, study treatment, and agrees not to donate eggs (ova, oocytes) to others or freeze/store these for her own use for the purpose of reproduction during this period. The investigator should evaluate the potential for contraceptive method failure (i.e., noncompliance, recently initiated) in relationship to the first dose of study intervention.

   C. A WOCBP must have negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention.

   D. If a urine test cannot be confirmed as negative (i.e., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

   E. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
5. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered in combination with platinum doublet chemotherapy concomitantly as first line treatment. Participants who have received Anti-PD-1/PD-L1(either as monotherapy or in combination with chemotherapy) as initial treatment at early-stage or locally advanced NSCLC should NOT be enrolled in this study. Anti-PD-1/PD-L1 treatment progression is defined by meeting all of the following criteria:

   A. Has received at least 2 doses of an approved anti-PD-1/L1 mAb

   B. Has demonstrated disease progression after anti-PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression. Eligible participants should have at least 2 pre-study images as confirmed evidence of PD (assessed by investigator) on treatment of anti-PD-1/L1 mAb before the study intervention.

   C. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb,
6. Have confirmation that EGFR-, ALK-, or ROS1-directed therapy is not indicated as primary therapy. Subjects who have failed directed therapy are not eligible for the study.
7. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
8. Have measurable disease (at least 1 measurable lesion by CT or MRI) based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
10. Have a life expectancy of at least 3 months and adequate organ function as defined in the following table.
11. Have adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP≤150/90mmHg and no change in antihypertensive medications within 1 week before treatment initiation.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment initiation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy at any stage of disease with any anti-VEGF-TKIs (i.e. Bevacizumab, Lenvatinib, Anlotinib, Apatinib, etc.) as monotherapy or in combination with an anti-PD-1/L1 inhibitor.
3. Has received prior Paclitaxel, Docetaxel or Albumin-paclitaxel as monotherapy or in combination with other therapies at any stage of disease.
4. Has received prior radiotherapy within 2 weeks of start of study intervention or has received lung radiation therapy >30 Gy within 6 months before the first dose of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has had major surgery within 3 weeks prior to first dose of study interventions.

   Note: Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility.
6. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
7. Has radiographic evidence of major blood vessel invasion/infiltration. In the chest, major blood vessels include the main pulmonary artery, the left and right pulmonary arteries, the 4 major pulmonary veins, the superior or inferior vena cava, and the aorta.

   Note: The degree of proximity to major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
8. Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.
9. Has urine protein ≥1 g/24 hours. Note: Participants with proteinuria ≥2+ (≥100 mg/dL) on urine dipstick testing or urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria.
10. Has a LVEF below the institutional (or local laboratory) normal range, as determined by echocardiogram (ECHO). OR has Prolongation of QTcF interval to >480 ms according to ECG.
11. Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
12. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
13. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
14. Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.

    Note: Medically controlled arrhythmia would be permitted.
15. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
16. Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of disease recurrence for 3 years since initiation of that therapy. Note: The requirement for no evidence of disease for 3 years does not apply to the NSCLC for which a participant is enrolled in the study. This time requirement also does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
17. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
18. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
19. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
20. Has an active infection requiring systemic therapy.
21. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
22. Has a sensitivity to any of the excipients contained in Albumin-paclitaxel and/or Lenvatinib.
23. Has a known history of Human Immunodeficiency Virus (HIV) infection.
24. Has active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) or Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by local health authority
25. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
26. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
27. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
28. Has had an allogenic tissue/solid organ transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | About 18 months
  Objective response rate (ORR) assessed per the Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Overall survival | About 36 months
  Overall survival (OS)
Progression-free survival | About 24 months
  Progression-free survival (PFS) assessed per RECIST v1.1
Duration of response | About 24 months
  Duration of response (DoR) assessed per RECIST v1.1
Treatment-related adverse events | About 24 months
  Treatment-related adverse events (TRAEs) assessed by CTCAE v5.0

OTHER OUTCOMES:
Single cell sequencing of tumor specimens | About 36 months
  Tumor specimens were collected before and after treatment for single cell assays to assess changes in the tumor immune microenvironment

CONTACTS AND LOCATIONS:
Overall Officials: Shikai Wu, Principal Investigator — Peking Univerisity First Hospital
Locations (1):
- Peking University First Hospital Ethics Committee, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No